CLINICAL TRIAL: NCT03802578
Title: The Impact of Exercise on Hand Function, on Activities of Daily Living (ADLs) Performance and Quality of Life of Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: The Impact of Exercise on Hand Function, Daily Activities Performance and Quality of Life of SLE' Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Maria Tektonidou, Ass. Professor Medical School, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 680/10-06-2016
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus; Arthralgia
Keywords: Exercise; Hand function; Quality of Life
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthralgia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXERCISE GROUP (Experimental): Patients in the exercise group performed a program of strengthening, stretching and resistance upper limbs exercises (Hand exercise), of 30 minutes duration daily, for 12 weeks in addition to medical care.
  Interventions: Behavioral: HAND EXERCISE
- CONTROL GROUP (No Intervention): Patients in the control group continued their usual medical care.

INTERVENTIONS:
Behavioral: HAND EXERCISE
  Arms: EXERCISE GROUP

SUMMARY:
A total of 240 consecutive SLE patients fulfilling the SLICC classification criteria was evaluated. Sixty two patients who met the inclusion criteria were randomly assigned to the exercise group (n=32) or the control group (n=30).

Patients in the exercise group performed a program of strengthening, stretching and resistance upper limbs exercises, of 30 minutes duration daily, for 12 weeks. Performance of daily activities was evaluated with the DASH and HAQ questionnaires, grip and pinch strength with the Jamar dynamometer and pinch gauge tools respectively, dexterity with the Purdue pegboard test and the quality of life with the LUPUSQoL questionnaire at 0, 6, 12 (end of the exercise program) and 24 weeks for both groups. SLE activity and cumulative organ damage were evaluated with the SLE disease activity index 2000 (SLEDAI-2K) and SLICC/ACR-DI, respectively.

DETAILED DESCRIPTION:
A total of 240 consecutive SLE patients fulfilling the SLICC classification criteria was evaluated. Sixty two patients who met the inclusion criteria [age>18, upper limb arthralgias, and DASH (Disabilities of the Arm, Shoulder, and Hand) questionnaire score>10)] were randomly assigned to the exercise group (n=32) or the control group (n=30).

Patients in the exercise group performed a program of strengthening, stretching and resistance upper limbs exercises, of 30 minutes duration daily, for 12 weeks. Performance of daily activities was evaluated with the DASH and HAQ questionnaires, grip and pinch strength with the Jamar dynamometer and pinch gauge tools respectively, dexterity with the Purdue pegboard test and the quality of life with the LUPUSQoL questionnaire at 0, 6, 12 (end of the exercise program) and 24 weeks for both groups. SLE activity and cumulative organ damage were evaluated with the SLE disease activity index 2000 (SLEDAI-2K) and SLICC/ACR-DI, respectively.

ELIGIBILITY:
Inclusion Criteria:

* SLE patients fulfilling the SLICC classification criteria
* Upper limb arthralgias
* DASH score>10
* Stable drug regimen≥3 months

Exclusion Criteria:

* Hand fracture or surgery in last 6 months
* Physiotherapy program in last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
change of DASH questionnaire | Baseline, 6, 12, 24 weeks
  Hand function was measured with DASH Questionnaire

SECONDARY OUTCOMES:
change of HAQ questionnaire | Baseline, 6, 12, 24 weeks
  Hand function was measured with HAQ Questionnaire
change of Grip strength | Baseline, 6, 12, 24 weeks
  Grip strength was measured with Jamar Dynamometer
change of Pinch strength | Baseline, 6, 12, 24 weeks
  Pinch strength was measured with Jamar pinch gauge
change of Dexterity | Baseline, 6, 12, 24 weeks
  Dexterity was measured with Purdue Pegboard test
change of Quality of Life | Baseline, 6, 12, 24 weeks
  Quality of Life was measured with LupusQoL Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: MARIA TEKTONIDOU, Ass. Prof, Principal Investigator — National and Kapodistrian University of Athens
Locations (2):
- Greece (2):
  - General Hospital of Athens 'Laiko', Athens, Attica
  - General Hospital of Elefsina 'Thriasio', Elefsina, Attica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keramiotou K, Anagnostou C, Kataxaki E, Galanos A, Sfikakis PP, Tektonidou MG. The impact of upper limb exercise on function, daily activities and quality of life in systemic lupus erythematosus: a pilot randomised controlled trial. RMD Open. 2020 Jan;6(1):e001141. doi: 10.1136/rmdopen-2019-001141. PMID 31958285